CLINICAL TRIAL: NCT01482572
Title: Feasibility of Gene Expression Profiling Using Low-volume Lung Aspirate
Brief Title: Feasibility of Mutational Analysis of Non-Small Cell Lung Cancer (NSCLC) Using Low-volume Lung Aspirates
Status: Withdrawn | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-10-078
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Lung Cancer
Keywords: biopsy; needle aspiration; mutational analysis
MeSH Terms: conditions — Lung Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lung tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Gene profiling Success
  Interventions: Procedure: biopsy

INTERVENTIONS:
Procedure: biopsy — percutaneous lung biopsy and aspiration

SUMMARY:
The purpose of this study is to evaluate the feasibility of aspiration samples for mutational analysis in patients with a non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
The investigators will compare results of mutational analysis from a core needle biopsy and fine needle aspiration.

ELIGIBILITY:
Inclusion Criteria:

* primary tumor or a metastatic lung lesion requested for mutational analysis

Exclusion Criteria:

* a) lesions located adjacent to the large central bronchi or vessels
* b) peribronchovascular lesions with prominent internal CT air-bronchograms, which were considered difficult to be avoided by needle pass
* c) lesions in patient with severe respiratory compromise

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Success rates for mutation analysis | one year

SECONDARY OUTCOMES:
Technical success rate of biopsy procedure | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ho Yun Lee, Dr., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea